CLINICAL TRIAL: NCT00408395
Title: A Phase II, Observer-Blind, Randomized, Parallel Groups, Multicenter, Exploratory Clinical Study to Evaluate the Immunogenicity and Safety of One and Two 0.25 mL Intramuscular Doses of a Commercially Available Influenza Vaccine Versus Two 0.25 mL Intramuscular Doses of a Commercially Available Influenza Vaccine in Healthy Children
Brief Title: Safety and Immunogenicity of 2 Commercially Available Influenza Vaccines in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70P2; 2006-003181-34
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-12

CONDITIONS: Influenza
Keywords: influenza; children; vaccine; influenza disease
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1: Trivalent Seasonal Influenza Vaccine (Experimental)
  Interventions: Biological: Influenza vaccine
- 2: Adjuvanted Trivalent Seasonal Influenza Vaccine (Experimental)
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Seasonal Influenza Vaccine

SUMMARY:
This is a study of the safety and immunogenicity of three commercially available influenza vaccines in children.

DETAILED DESCRIPTION:
A Phase II, Observer-Blind, Randomized, Parallel Groups, Multicenter, Exploratory Clinical Study to Evaluate the Immunogenicity and Safety of One and Two 0.25 mL Intramuscular Doses of a commercially available influenza vaccine versus Two 0.25 mL Intramuscular Doses of a commercially available influenza vaccine in Healthy Children

ELIGIBILITY:
Inclusion Criteria:

* 6 months to < 36 months of age

Exclusion Criteria:

* Any severe acute respiratory disease and infections requiring systemic antibiotic or antiviral therapy ongoing or resolved within 30 days prior to study start (chronic antibiotic therapy for urinary tract prophylaxis is acceptable)
* Other serious diseases such as: cancer, autoimmune disease (including rheumatoid arthritis), diabetes mellitus, chronic pulmonary disease, acute or progressive hepatic or renal disease, or surgery planned during the study period.
* Known or suspected impairment/alteration of immune function
* History of hypersensitivity to any component of the study vaccine, egg products or other vaccine component, or impairment/alteration of immune function

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 281 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of the 2 vaccines in terms of post-immunization geometric mean titers (GMTs), as measured by the hemagglutination inhibition (HI) test

SECONDARY OUTCOMES:
To evaluate the immunogenicity of the 2 vaccines in terms of seroprotection, and seroconversion or significant increase, as measured by HI test
To evaluate the safety and tolerability of the 2 vaccines administered 4 weeks apart

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines (formerly Chiron Vaccines), Study Chair — Novartis
Locations (1):
- University of Tampere Medical School, Tampere, Finland

REFERENCES:
- [Result] Vesikari T, Pellegrini M, Karvonen A, Groth N, Borkowski A, O'Hagan DT, Podda A. Enhanced immunogenicity of seasonal influenza vaccines in young children using MF59 adjuvant. Pediatr Infect Dis J. 2009 Jul;28(7):563-71. doi: 10.1097/INF.0b013e31819d6394. PMID 19561422